CLINICAL TRIAL: NCT06150534
Title: Evaluating the Treatment Experience During Initiation of Subcutaneous Immunoglobulin Replacement (SCIG) Therapy at Home Using Alexa Skill
Brief Title: At-Home Subcutaneous Immunoglobulin Replacement Therapy Using Alexa Skill
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: PID-5005
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: Drug Therapy
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult Patients with PID: Adult patients with PID who recently started or will soon begin to complete SCIG (HyQvia or Cuvitru) infusions independently will be interviewed before and/or after the use of Alexa Skill.
  Interventions: Other: No Intervention
- Caregivers of Patients with a Self-reported Diagnosis of PID: Caregivers who recently started or will soon begin infusing SCIG (HyQvia or Cuvitru) for patients with a self-reported diagnosis of PID will be interviewed before and/or after the use of Alexa Skill.
  Interventions: Other: No Intervention
- Healthcare Professionals (HCPs): HCPs, specifically, clinical immunologists who prescribe SCIG for the treatment of PID and nurses who have experience administering SCIG will be interviewed after the use of Alexa Skill.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to determine the impact of digital health technology, such as Alexa Skill, used to support the initiation of home-based subcutaneous immunoglobulin (SCIG) treatment, treatment management, and overall participant experience.

DETAILED DESCRIPTION:
This is a non-interventional, observational study to identify relevant concepts of SCIG treatment experience, as well as satisfaction regarding Alexa skill-assisted SCIG initiation, infusion, and disease/therapy management.

The study will enroll approximately 36 participants (26 patients/caregivers and 10 healthcare professionals [HCPs]). Participants will be enrolled into following observational Cohorts:

* Adult patients with primary immunodeficiency (PID)
* Caregivers of patients with a self-reported diagnosis of PID
* HCPs who prescribe SCIG for patients with PID

Interviews will be conducted by a trained qualitative research interviewer with patients, caregivers, and HCPs, and self-reported data will be collected.

This trial will be conducted in the United States. The overall duration of the study will be approximately 4 months.

ELIGIBILITY:
Inclusion Criteria:

Patients and caregivers:

* Adult patient (aged 18 years or older) with PID who recently initiated (within 4 months) or will soon initiate (within 30 days) HyQvia or Cuvitru at home or caregiver (aged 18 years or older) supporting participants (any age) with PID who recently initiated (within 4 months) or will soon initiate (within 30 days) HyQvia or Cuvitru at home.
* Patient has a self-reported physician diagnosis of PID.
* Resides in the US or US territories.
* Can speak and read English fluently.
* Able to participate in an interview(s).
* Must have a wireless network (Wi-Fi) at home (cannot be a wireless hotspot).
* Must have an existing Amazon account.
* Must be willing to receive an Amazon Echo Show device and connect the device to Wi-Fi.
* Must have a smartphone and be willing to download and use the Alexa application to access the Alexa Skill test.

Additional criteria for patients and caregivers completing qualitative debriefing interviews:

* Must have at least 2 SCIG infusions (HyQvia or Cuvitru) at a residential home or residential assisted living facility within 6 to12 weeks.
* Must attest to use of Alexa Skill to support at-home SCIG infusions.

For HCPs:

* Resides in the US or US territories.
* Must be an immunologist or registered nurse/nurse practitioner.
* Licensed to practice in the US.
* Can speak and read English fluently.
* Able to participate in a debriefing interview.
* Willing to provide informed consent.
* Must have a wireless network (Wi-Fi).
* Must have an existing Amazon account.
* Must be willing to receive an Amazon Echo Show device and connect the device to Wi-Fi.
* Must have a smartphone and be willing to download and use the Alexa application to access the Alexa Skill test.
* Must attest to exploration of Alexa Skill as a support tool for patients and caregivers administering SCIG infusions at home.

Exclusion Criteria

• Patients who were previously on SCIG and transitioned to either HyQvia or Cuvitru SCIG product will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients and/or caregivers supporting patients with PID and HCPs involved in treating patients with PID who reside in the United States (US).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Identify Participant Experience, Including Convenience and Satisfaction, With Alexa Skill | 4 months
  Qualitative interviews with patients, caregivers, and HCPs who will be using the Alexa Skill to support initiation of SCIG for PID to characterize their experience, including convenience and satisfaction. Qualitative interviews will be semi-structured to comprehensively assess confidence and satisfaction, but also open-ended to give patients, families, and HCPs freedom to discuss their experience.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Research Triangle Park, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/122e9b02747d4a29?idFilter=%5B%22PID-5005%22%5D